CLINICAL TRIAL: NCT03174561
Title: Clinical Assessment of the Benefits of the Combination Inuline, Choline and Silymarin in Mitigating the Symptomatology in Patients With Irritable Bowel Syndrome
Brief Title: Inuline Supplement in Patients With Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: SC Fiterman Pharma SRL (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: STCL009
Record Dates: First submitted 2017-05-31; First posted 2017-06-02 (Actual); Last update posted 2017-06-02 (Actual); Status verified 2017-05

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Choline; Silymarin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inuline, Choline and Silymarin + Diet (Other): Patients diagnosed with Irritable bowel syndrome who will follow diet restrictions together with a dietary supplement.
  Intervention: Dietary Supplement, a combination of Inuline, Silymarin and Choline The dose: 1 sachet first 7 days and 1 sachet x 2 times daily for the next 21 days
  Interventions: Dietary Supplement: Inuline, Choline and Silymarin
- Diet restriction (Other): Patients diagnosed with Irritable bowel syndrome who will follow diet restrictions for 28 days. After the first month the patients are crossed between groups.
  Interventions: Other: diet restriction

INTERVENTIONS:
Dietary Supplement: Inuline, Choline and Silymarin — Combination of one sachet: Inuline (5000 mg), Silybum marianum seed extract (50 mg), Choline (37 mg) The dose: 1 sachet first 7 days and 1 sachet x 2 times daily for the next 21 days. Diet restriction is consider together with dietary supplement intake.
  Other Names: Stoptoxin plicuri
  Arms: Inuline, Choline and Silymarin + Diet
Other: diet restriction — diet restriction for 28 days
  Arms: Diet restriction

SUMMARY:
The study investigate the efficacy of the combination inuline, choline and silymarin in alleviating the symptomatology of the patients with irritable bowel syndrome with constipation in a randomized, cross-over, no treatment controlled study.

DETAILED DESCRIPTION:
In this study patients diagnosed using Rome IV criteria with irritable bowel syndrome with constipation are included. The study was approved by the Ethic Committee of the University of Medicine and Pharmacy "Gr. T Popa" Iasi to be conducted at the Institute of Gastroenterology and Hepatology of Clinical Emergency Hospital "Sf. Spiridon" Iasi. The patients are assigned after a randomized scheme to one of the groups: diet restriction scheme or diet restriction scheme plus a product with inuline, choline and silymarin. After 28 days the patients are crossed between the groups and followed for additional 28 days diet scheme with or without inuline, choline and silymarin supplementation. All the patients are evaluated initially, in the day 28 and in the day 57 for the stool habits, stool characteristics using Brystol Scale and symptoms severity (abdominal pain, frequency of abdominal pain, bloating severity, patients satisfaction in relation with stool frequency and the impact of IBS on daily activity) as appreciated by the patients for the last 10 days.

The acquired data will be analyzed and published.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-75 years, diagnosed with Irritable Bowel Syndrome using Roma IV criteria

Exclusion Criteria:

* Patients with IBS with predominant diarrhea or mixt symptoms
* Patients with known hypersensitivity to any of the ingredients of the dietary supplement
* Patients who used prebiotic, probiotic or laxative products in the last 10 days
* Pregnancy and lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2018-02-28 (Estimated); Study Completion 2018-04-30 (Estimated)

PRIMARY OUTCOMES:
IBS symptoms severity score | the last 10 days
  visual analogue scale for IBS symptoms severity will be used
number of bowel movements | the last 7 days
  number of bowel movements/week

CONTACTS AND LOCATIONS:
Overall Officials: Vasile L Drug, Lecturer, Principal Investigator — Institute of Gastroenterology and Hepatology of Clinical Emergency Hospital "Sf. Spiridon" Iasi; Ioan Chirila, Consultant, Study Chair — National Institute of public Health
Locations (1):
- Institute of Gastroenterology and Hepatology of Clinical Emergency Hospital "Sf. Spiridon", Iași, Romania

IPD SHARING:
Plan to Share IPD: No